CLINICAL TRIAL: NCT04490187
Title: tDCS and Motor Learning in Children With DCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Jill Zwicker, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H17-02513
Record Dates: First submitted 2020-01-18; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Developmental Coordination Disorder
Keywords: motor skills disorders; tDCS; task-specific intervention; occupational therapy
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: Children with DCD with be recruited and randomized to receive active stimulation or sham tDCS
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to sham vs active stimulation groups. The outcomes assessor will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS stimulation (Experimental): tDCS will be applied over the left motor cortex at 1 mA for 30 min. The current will be ramped up to 1 mA over 45-60 s, held for 30 min, and ramped down to 0 mA over 45-60 s.
  Interventions: Behavioral: Motor Learning
- Sham tDCS stimulation (Sham Comparator): tDCS will be ramped up and held for only 60 s before it is slowly ramped down. This procedure, called the Fade-in-Short Stimulation-Fade out, has shown its reliability as an effective sham technique through making the same tolerability and transient scalp sensation as active stimulation in both adults (Ambrus 2012) and children (Ciechanski 2017).
  Interventions: Behavioral: Motor Learning

INTERVENTIONS:
Behavioral: Motor Learning — Over three consecutive days, each child will perform five blocks of Purdue Pegboard Test: one block before, three blocks during, and one block after tDCS. Each block consists of three repetitions of Purdue Pegboard Test with the right hand. The children have to place pins into a pegboard as fast as they can in 30 seconds. It will take up to 10 minutes of brain stimulation time.
  After the Purdue Pegboard Test, each child will receive cognitive-based intervention for printing skills for 20 minutes while receiving tDCS. "Printing Like a Pro!" (Montgomery 2017) -a cognitive approach to teaching printing to primary school-age children-will be used to teach letters which each child has the most difficulty printing legibly as identified on a formal assessment of handwriting-ETCH (manuscript) (Amundson 1995).

SUMMARY:
Children with a neurodevelopmental condition called developmental coordination disorder (DCD) struggle to learn motor skills and perform daily activities, such as tying shoelaces, printing, riding a bicycle, or playing sports. Evidence suggests that motor-based interventions combined with non-invasive brain stimulation to the motor cortex (transcranial direct-current stimulation, tDCS) has been effective in improving motor skills in children with cerebral palsy and other neurodevelopmental disorders, but few studies have examined tDCS in chidlren with DCD. The purpose of this randomized, blinded, sham-controlled interventional trial is to explore the effectiveness of anodal tDCS over M1 combined with a motor learning task in increasing motor skill learning in children with DCD.

DETAILED DESCRIPTION:
Transcranial direct-current stimulation (tDCS) is one of the most common non-invasive brain stimulation techniques but applications in pediatric populations are relatively unexplored. tDCS applies a weak electric current over the scalp to modulate cortical excitability. Anodal stimulation excites the stimulated brain region. Anodal tDCS applied to the motor cortex contralateral to the trained hand enhances motor learning across single or multiple day training sessions (Reis 2009). tDCS has shown promising effects in the developing brain including the potential to enhance motor skills that may then be transferred to other untrained skills in typically developing children (Ciechanski 2017). tDCS is safe and tolerable and a feasible technique with only mild short-term adverse effects (e.g., redness, tingling, itching, and burning sensation) in children. The adverse effects usually occur at electrode sites and disappear within a few minutes after stimulation starts (Krishnan 2015).

Combined with motor-based interventions, tDCS can enhance motor performance in adults (Reis 2009, 2011) and children (Gillick 2014; Grecco 2017; Kirton 2017; Moura 2016). It is currently being used in combination with other treatments (e.g., behavioural therapy and neurorehabilitation) in children and adolescents with neurodevelopmental disorders (Muszkat 2016), including Autism Spectrum Disorder (Amatachaya 2014) and Attention-Deficit/Hyperactivity Disorder (ADHD) (Bandeira 2016), as well as motor disorders such as Cerebral Palsy (Gillick 2014; Grecco 2017; Kirton 2017; Moura 2016). However, the effect of tDCS on skill motor learning in children with Developmental Coordination Disorder (DCD) is largely unexplored.

DCD is a chronic motor disorder of unknown etiology that affects 5-6% of school-aged children in Canada (APA, 2013). DCD interferes with children's academic achievement and limits their ability to participate in daily activities (e.g., printing, getting dressed, tying their shoes, riding a bike, using cutlery), as well as vocational activities, leisure, and play (APA, 2013).15 Subsequently, children may develop psychosocial difficulties, including low self-esteem, depression, anxiety, loneliness, problems with peers, and poor participation in physical and social activities (Zwicker 2013). DCD is a lifelong condition, and 75% of children with DCD will continue to experience motor difficulties as adults if they don't receive proper treatment (Kirby 2014). Up to half of children with DCD also have co-occurring ADHD (Piek 1999).

Several brain regions have been implicated in DCD, including the cerebellum, basal ganglia, parietal lobe, and parts of the frontal lobe (e.g., dorsolateral prefrontal cortex or DLPFC) (Biotteau 2016). The primary motor cortex (M1) is located in the dorsal part of the frontal lobe and is functionally connected to other motor areas. However, the functional connectivity between M1 and brain regions involved in motor functioning and sensorimotor processing, such as striatum and angular gyrus, may be decreased in children with DCD (McLeod 2014). Targeting such specific brain regions in rehabilitation might be effective in improving the motor outcomes of affected children.

Currently, the most beneficial interventions to improve the motor performance of children with DCD are task-oriented approaches that focus on learning a particular task rather than on the body functions required to perform a task (Smits-Engelsman 2013). A number of task-oriented approaches are commonly used to treat children with DCD (Niemeijer 2007; Polatajko 2001). The investigators believe that brain stimulation can enhance motor learning and the effect of task-oriented approaches in children with DCD. To better understand tDCS as a treatment for children with DCD, as the first step, it is critical to investigate whether tDCS can enhance motor skill learning in this population. Therefore, the investigators aim to conduct a randomized, blinded, sham-controlled interventional trial of anodal tDCS over M1 combined with a motor learning task to assess its effectiveness on motor skill learning in children with DCD. This is a pilot study to determine a sample size for a larger study.

AIMS AND HYPOTHESES

Aim 1: To determine if transcranial direct current stimulation (tDCS) enhances motor learning in children with DCD.

Hypothesis 1: Compared to children in sham group, children in stimulation group will show better functional outcomes faster motor learning in each session (online learning) and after 3 sessions.

Aim 2: To determine the longevity of tDCS effects on motor learning in children with DCD.

Hypothesis 2: Children in stimulation group will maintain their motor learning after 6 weeks compared to the sham group.

METHODOLOGY

Study Design: This study is a randomized, sham-controlled, double-blinded trial. Participants will be randomly assigned to active or sham stimulation.

Participants: Children will be recruited from established cohorts of children with DCD who were assessed at BC Children's Hospital or Sunny Hill Health Centre for Children (Vancouver, BC) and who meet DSM-5 diagnostic criteria (American Psychiatric Association, 2013).

Sample size: Sample size was calculated based on a randomized sham-control designed study in typically-developing children receiving M1 A-tDCS or sham tDCS over 3 consecutive days of Purdue Pegboard Test training.4 Sample size calculation suggested a total of 14 subjects, 7 subjects per group, would have a power of 95% to detect improvement in Purdue Pegboard Test (effect size = 2.58) with a type-1 error of 0.05.

Procedure: After screening and recruitment, parents will consent and children will assent to take part in the study. We will randomize children to active or sham stimulation groups; a statistician will randomize participants using computer-generated sequential blocks of 4 to 6. Randomization codes will be kept in sealed opaque envelopes until study enrollment. A research graduate student with training in occupational therapy will be blinded to group assignments and will assess children using Purdue Pegboard Test (PPT; Tiffin 1968), Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2; Bruininks 2005), and Evaluation Tool of Children's Handwriting (ETCH; Amundson, 1995). Then, children will receive 3 days of tDCS for 30 minutes each day; during the first 10 minutes, children will complete Purdue Pegboard Test Training (to assess learning of a motor task), followed by 20 minutes of handwriting practice using "Printing Like a Pro!"(Montgomery 2017), to assess learning of a functional motor task). An occupational therapist will re-assess the children at the end of the last day of training and again 6 weeks later.

Interventions

tDCS: Direct current will be delivered using a transcranial electrical stimulator approved by Health Canada (Soterix Medical Inc., New York, USA) (Soterix Medical, 2016). Stimulation will be applied to the scalp through two 5×7 cm sponge saline-soaked electrodes: active and reference. A simple headgear system, including the EASYpads and EASYstraps, will hold the electrodes in place. In the active stimulation and sham groups, the anode (active electrode) will be positioned over the left primary motor cortex with the cathode (reference electrode) over right forehead in supraorbital area. The international 10/20 electroencephalography electrode system will be used to localize the M1 (Klem 1999). The dominant left motor cortex will be stimulated because the investigators aim to simultaneously train the dominant hand for a motor learning task and a functional task. The stimulation will be applied at 1 mA for 30 min. One mA of anodal stimulation may cause brain current densities in children on average comparable to densities seen in adults exposed to 2 mA current (Kessler 2013) and the subsequent excitability might last longer than one hour (Moliadze 2015). For active stimulation groups, the current will be ramped up to 1 mA over 45-60 s, held for 30 min, and ramped down to 0 mA over 45-60 s. For the sham groups, stimulation will be ramped up and held for only 60 s before it is slowly ramped down. This procedure, called the Fade-in-Short Stimulation-Fade out, has shown its reliability as an effective sham technique through making the same tolerability and transient scalp sensation as active stimulation in both adults (Ambrus 2012) and children (Ciechanski 2017). In case of any "Serious Adverse Events" (e.g., second-degree scalp burn at the site of electrode pad, or clinical seizure) occurring during the course of study, it will be stopped immediately.

Motor Learning Task: Over three consecutive days, each child will perform five blocks of Purdue Pegboard Test: one block before, three blocks during, and one block after tDCS. Each block consists of three repetitions of Purdue Pegboard Test with the right hand. The children have to place pins into a pegboard as fast as they can in 30 seconds. It will take up to 10 minutes of brain stimulation time.

Functional Motor Task: After the Purdue Pegboard Test, each child will receive cognitive-based intervention for printing skills for 20 minutes while receiving tDCS. "Printing Like a Pro!" (Montgomery 2017) -a cognitive approach to teaching printing to primary school-age children-will be used to teach letters which each child has the most difficulty printing legibly as identified on a formal assessment of handwriting-ETCH (manuscript) (Amundson 1995).

Data Analysis Plan:

Purdue Pegboard Test is the primary outcome measure of interest. To measure online learning within one session and off-line learning across sessions, we will apply Repeated Measure Analysis of Co-variance (ANCOVA), with an α level of 0.05. To measure effect of intervention and retention, we will apply a paired t-test and Repeated Measure ANCOVA to the primary and secondary outcomes. Two-way ANCOVA and independent t-test will also be used to compare groups (stimulation versus sham). MABC-2 scores and attention level as assessed by Conner's ADHD Index will be used as covariates to account for individual differences in attention and motor skills.

Significance:

This is the first study of its kind to both investigate the effect of brain stimulation in motor learning in children with DCD and integrate technology to improve functional motor learning for children with DCD. This study will contribute to planning more effective interventions for these children to improve both their motor skills and functional outcomes. Additionally, findings will be of interest to pediatric clinicians (e.g., occupational therapists) and parents seeking more efficient approaches for these children, as well as researchers, students, and policy makers in the field of neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* a score of ≤5th percentile in Manual Dexterity composite of the Movement Assessment Battery for Children-2 (MABC-2), as we are focusing on fine motor tasks in the study (Henderson 2007)
* meet DCD criteria on the DCD Questionnaire (Wilson 2007)
* right-handed as per the Edinburg Handedness Inventory (Oldfield 1971)

Exclusion Criteria:

* born preterm (gestation week<37 weeks)
* diagnosed with any other neurodevelopmental disability such as Autism Spectrum Disorder (except ADHD)
* history of any neurological disorders
* taking any neuropsychiatric medications
* history of migraines
* having a scalp or skin condition (e.g., psoriasis or eczema)
* having a metallic implants (e.g., surgical clips or pacemaker)
* history of seizure or epilepsy

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Purdue Pegboard Test (Tiffin 1968) | Before and after intervention; 6 weeks after intervention
  A standardized assessment that measures manual dexterity and bilateral coordination¬-the participants have 30 seconds to place pins into pegboard using their (1) right hand, (2) left hand, and (3) both hands, as well as another 30 seconds to assemble pins, washers and collars with both hands.

SECONDARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2: Bruininks 2005) fine motor composite | Before and after intervention; 6 weeks after intervention
  Assesses fine motor precision, fine motor integration, and manual dexterity. Scores are reported as a percentile rank; higher scores indicate better fine motor skills.
Evaluation Tool of Children's Handwriting (ETCH: Amundson 1995) | Before and after intervention; 6 weeks after intervention
  Assesses children's legibility and speed of writing lower-case letters in manuscript

OTHER OUTCOMES:
Conner's ADHD Index (Conners 2009) | Before intervention
  parent report of children's symptoms of inattention and hyperactivity to measure of attention as a co-variate in the analyses
tDCS Adverse Effects Questionnaire (Brunoni 2011) | After each session of tDCS stimulation (active or sham) - daily for 3 consecutive days
  Collect information regarding severity of symptoms immediately following tDCS. It screens symptoms including headache, neck pain, scalp pain, tingling, itching, burning sensation, skin redness, sleepiness, trouble concentrating, acute mood change, and any other self-reported symptoms. Higher score indicates more adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Jill G Zwicker, PhD, OT, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589
- [Background] Ciechanski P, Kirton A. Transcranial Direct-Current Stimulation Can Enhance Motor Learning in Children. Cereb Cortex. 2017 May 1;27(5):2758-2767. doi: 10.1093/cercor/bhw114. PMID 27166171
- [Background] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Background] Reis J, Fritsch B. Modulation of motor performance and motor learning by transcranial direct current stimulation. Curr Opin Neurol. 2011 Dec;24(6):590-6. doi: 10.1097/WCO.0b013e32834c3db0. PMID 21968548
- [Background] Gillick BT, Kirton A, Carmel JB, Minhas P, Bikson M. Pediatric stroke and transcranial direct current stimulation: methods for rational individualized dose optimization. Front Hum Neurosci. 2014 Sep 19;8:739. doi: 10.3389/fnhum.2014.00739. eCollection 2014. PMID 25285077
- [Background] Grecco LA, Oliveira CS, Duarte NA, Lima VL, Zanon N, Fregni F. Cerebellar transcranial direct current stimulation in children with ataxic cerebral palsy: A sham-controlled, crossover, pilot study. Dev Neurorehabil. 2017 Apr;20(3):142-148. doi: 10.3109/17518423.2016.1139639. Epub 2016 Mar 22. PMID 27003795
- [Background] Kirton A, Ciechanski P, Zewdie E, Andersen J, Nettel-Aguirre A, Carlson H, Carsolio L, Herrero M, Quigley J, Mineyko A, Hodge J, Hill M. Transcranial direct current stimulation for children with perinatal stroke and hemiparesis. Neurology. 2017 Jan 17;88(3):259-267. doi: 10.1212/WNL.0000000000003518. Epub 2016 Dec 7. PMID 27927938
- [Background] Moura RC, Santos CA, Grecco LA, Lazzari RD, Dumont AJ, Duarte NC, Braun LA, Lopes JB, Santos LA, Rodrigues EL, Albertini G, Cimolin V, Galli M, Oliveira CS. Transcranial direct current stimulation combined with upper limb functional training in children with spastic, hemiparetic cerebral palsy: study protocol for a randomized controlled trial. Trials. 2016 Aug 17;17(1):405. doi: 10.1186/s13063-016-1534-7. PMID 27530758
- [Background] Muszkat D, Polanczyk GV, Dias TG, Brunoni AR. Transcranial Direct Current Stimulation in Child and Adolescent Psychiatry. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):590-7. doi: 10.1089/cap.2015.0172. Epub 2016 Mar 30. PMID 27027666
- [Background] Amatachaya A, Auvichayapat N, Patjanasoontorn N, Suphakunpinyo C, Ngernyam N, Aree-Uea B, Keeratitanont K, Auvichayapat P. Effect of anodal transcranial direct current stimulation on autism: a randomized double-blind crossover trial. Behav Neurol. 2014;2014:173073. doi: 10.1155/2014/173073. Epub 2014 Oct 30. PMID 25530675
- [Background] Bandeira ID, Guimaraes RS, Jagersbacher JG, Barretto TL, de Jesus-Silva JR, Santos SN, Argollo N, Lucena R. Transcranial Direct Current Stimulation in Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD): A Pilot Study. J Child Neurol. 2016 Jun;31(7):918-24. doi: 10.1177/0883073816630083. Epub 2016 Feb 15. PMID 26879095
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders - 5th ed. (DSM-5). Washington, DC: American Psychiatric Association; 2013.
- [Background] Zwicker JG, Harris SR, Klassen AF. Quality of life domains affected in children with developmental coordination disorder: a systematic review. Child Care Health Dev. 2013 Jul;39(4):562-80. doi: 10.1111/j.1365-2214.2012.01379.x. Epub 2012 Apr 20. PMID 22515477
- [Background] Kirby A, Sugden D, Purcell C. Diagnosing developmental coordination disorders. Arch Dis Child. 2014 Mar;99(3):292-6. doi: 10.1136/archdischild-2012-303569. Epub 2013 Nov 19. PMID 24255567
- [Background] Piek JP, Pitcher TM, Hay DA. Motor coordination and kinaesthesis in boys with attention deficit-hyperactivity disorder. Dev Med Child Neurol. 1999 Mar;41(3):159-65. doi: 10.1017/s0012162299000341. PMID 10210248
- [Background] Biotteau M, Chaix Y, Blais M, Tallet J, Peran P, Albaret JM. Neural Signature of DCD: A Critical Review of MRI Neuroimaging Studies. Front Neurol. 2016 Dec 16;7:227. doi: 10.3389/fneur.2016.00227. eCollection 2016. PMID 28018285
- [Background] McLeod KR, Langevin LM, Goodyear BG, Dewey D. Functional connectivity of neural motor networks is disrupted in children with developmental coordination disorder and attention-deficit/hyperactivity disorder. Neuroimage Clin. 2014 Mar 26;4:566-75. doi: 10.1016/j.nicl.2014.03.010. eCollection 2014. PMID 24818082
- [Background] Smits-Engelsman BC, Blank R, van der Kaay AC, Mosterd-van der Meijs R, Vlugt-van den Brand E, Polatajko HJ, Wilson PH. Efficacy of interventions to improve motor performance in children with developmental coordination disorder: a combined systematic review and meta-analysis. Dev Med Child Neurol. 2013 Mar;55(3):229-37. doi: 10.1111/dmcn.12008. Epub 2012 Oct 29. PMID 23106530
- [Background] Niemeijer AS, Smits-Engelsman BC, Schoemaker MM. Neuromotor task training for children with developmental coordination disorder: a controlled trial. Dev Med Child Neurol. 2007 Jun;49(6):406-11. doi: 10.1111/j.1469-8749.2007.00406.x. PMID 17518923
- [Background] Polatajko HJ, Mandich AD, Miller LT, Macnab JJ. Cognitive orientation to daily occupational performance (CO-OP): part II--the evidence. Phys Occup Ther Pediatr. 2001;20(2-3):83-106. PMID 11345514
- [Background] Henderson SE, Sugden DA, Barnett AL. Movement Assessment Battery for Children - 2nd ed. Psychological Corporation London; 2007.
- [Background] Wilson, B.N., Kaplan, B.J., Crawford, S.G., & Roberts, G. (2007). Developmental Coordination Questionnaire 2007 (DCDQ'07). Available at:http://www.dcdq.ca.
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Conners CK. (2009). Conners3rd Edition (Conners 3). Toronto, ON: Multi-HealthSystems.
- [Background] Tiffin J. Purdue pegboard test. Chicago: Scientific Research Associates. 1968.
- [Background] Bruininks, R., & Bruininks, B. Bruininks-oseretsky test of motor proficiency. 2nd ed. Minneapolis, MN: NCS Pearson; 2005.
- [Background] Montgomery, I. & Zwicker, J.G. Printing like a pro! http://www.childdevelopment.ca/Libraries/Handwriting/Printing_Like_a_Pro_-_For_School_Staff.sflb.ashx
- [Background] Amundson, S. (1995). Evaluation tool of children's handwriting. Homer, AL: OT KIDS.
- [Background] Soterix Medical. Soterix medical launches PainX tDCS treatment in canada with health canada approval. https://soterixmedical.com/newsroom/press/2016/09/soterix-medical-launches-painx-tdcs-treatment-in-canada/26.
- [Background] Klem GH, Luders HO, Jasper HH, Elger C. The ten-twenty electrode system of the International Federation. The International Federation of Clinical Neurophysiology. Electroencephalogr Clin Neurophysiol Suppl. 1999;52:3-6. No abstract available. PMID 10590970
- [Background] Kessler SK, Minhas P, Woods AJ, Rosen A, Gorman C, Bikson M. Dosage considerations for transcranial direct current stimulation in children: a computational modeling study. PLoS One. 2013 Sep 27;8(9):e76112. doi: 10.1371/journal.pone.0076112. eCollection 2013. PMID 24086698
- [Background] Moliadze V, Schmanke T, Andreas S, Lyzhko E, Freitag CM, Siniatchkin M. Stimulation intensities of transcranial direct current stimulation have to be adjusted in children and adolescents. Clin Neurophysiol. 2015 Jul;126(7):1392-9. doi: 10.1016/j.clinph.2014.10.142. Epub 2014 Oct 28. PMID 25468234
- [Background] Ambrus GG, Al-Moyed H, Chaieb L, Sarp L, Antal A, Paulus W. The fade-in--short stimulation--fade out approach to sham tDCS--reliable at 1 mA for naive and experienced subjects, but not investigators. Brain Stimul. 2012 Oct;5(4):499-504. doi: 10.1016/j.brs.2011.12.001. Epub 2012 Feb 22. PMID 22405745
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389